CLINICAL TRIAL: NCT00329459
Title: A Randomized, Double-blind, Single Migraine Attack, Placebo -Controlled, Patallel-group Multicenter Study to Evaluate the Efficacy and Tolerability or Trexima (Sumatriptan Succinate/Naproxen Sodium) Tablets vs Placebo When Administered During the Mild Pain Phase of Menstrual Migraine in Women With Dysmenorrhea
Brief Title: Treximet (Sumatriptan/Naproxen Sodium), Formerly Known as TREXIMA, for Menstrual Migraine in Women With Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRX105850
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Migraine Disorders
Keywords: menstrual migraine; headache; early intervention; dysmenorrhea
MeSH Terms: conditions — Migraine Disorders; Headache; Dysmenorrhea | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm 1 (Experimental): Treximet (sumatriptan/naproxen sodium)
  Interventions: Drug: sumatriptan succinate/naproxen sodium
- arm 2 (Placebo Comparator): placebo to match
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sumatriptan succinate/naproxen sodium
  Arms: arm 1
Drug: placebo — placebo to match
  Arms: arm 2

SUMMARY:
This study was designed to determine efficacy of TREXIMA compared to placebo for the treatment of a menstrual migraine.

DETAILED DESCRIPTION:
A randomized, double-blind, single migraine attack, placebo-controlled, parallel group, multicenter study to evaluate the efficacy and tolerability of TREXIMA* (sumatriptan succinate/naproxen sodium) tablets vs placebo when administered during the mild pain phase of menstrual migraine in women with dysmenorrhea. (TREXIMET was formerly known as TREXIMA)

ELIGIBILITY:
Inclusion Criteria:

* At least a 6 month history of physician diagnosed migraine and typically experiences 2-6 migraine attacks per month.
* Typically experiences moderate to severe migraine pain preceded by a mild pain phase.
* Differentiate between mild migraine pain and other headache types.
* Women of childbearing potential must be on adequate contraception.

Exclusion Criteria:

* Pregnant and/or nursing mother.
* History of cardiovascular disease.
* Uncontrolled hypertension.
* Basilar or Hemiplegic migraine.
* History of stroke or transient ischemic attacks (TIA).
* History of epilepsy or treated with anti-epileptics within past 5 years.
* Impaired hepatic or renal function.
* History of gastrointestinal bleeding or ulceration.
* Allergy or hypersensitivity to aspirin or any other NSAID.
* Allergy or hypersensitivity to triptans.
* Participated in an investigational drug trial in the previous 4 weeks.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Score on a 4-point migraine pain scale for a single menstrual migraine attack | 2 to 48 hours

SECONDARY OUTCOMES:
Freedom from all migraine pain and symptoms, satisfaction, presence or absence of neck pain/discomfort, sinus pain/pressure, menstrual symptoms, recurrence of head pain, safety and tolerability | from 2 to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- United States (34):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fair Oaks, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Moorestown, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Plainview, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Independence, Ohio
  - GSK Investigational Site, Westerville, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Durham PL, Vause CV, Derosier F, McDonald S, Cady R, Martin V. Changes in salivary prostaglandin levels during menstrual migraine with associated dysmenorrhea. Headache. 2010 May;50(5):844-51. doi: 10.1111/j.1526-4610.2010.01657.x. Epub 2010 Mar 26. PMID 20353434
- [Result] Mannix LK, Martin VT, Cady RK, Diamond ML, Lener SE, White JD, Derosier FJ, McDonald SA. Combination treatment for menstrual migraine and dysmenorrhea using sumatriptan-naproxen: two randomized controlled trials. Obstet Gynecol. 2009 Jul;114(1):106-113. doi: 10.1097/AOG.0b013e3181a98e4d. PMID 19546766
- [Derived] Martin VT, Ballard J, Diamond MP, Mannix LK, Derosier FJ, Lener SE, Krishen A, McDonald SA. Relief of menstrual symptoms and migraine with a single-tablet formulation of sumatriptan and naproxen sodium. J Womens Health (Larchmt). 2014 May;23(5):389-96. doi: 10.1089/jwh.2013.4577. Epub 2014 Feb 28. PMID 24579886
- [Derived] Cady RK, Diamond ML, Diamond MP, Ballard JE, Lener ME, Dorner DP, Derosier FJ, McDonald SA, White J, Runken MC. Sumatriptan-naproxen sodium for menstrual migraine and dysmenorrhea: satisfaction, productivity, and functional disability outcomes. Headache. 2011 May;51(5):664-73. doi: 10.1111/j.1526-4610.2011.01894.x. PMID 21521204
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: TRX105850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: TRX105850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TRX105850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TRX105850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TRX105850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TRX105850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: TRX105850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register